CLINICAL TRIAL: NCT04577014
Title: A Multi-cohort Study of Retifanlimab With or Without Gemcitabine and Docetaxel in Patients With Advanced Sarcoma
Brief Title: Retifanlimab (Anti-PD-1 Antibody) With Gemcitabine and Docetaxel in Patients With Advanced Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-316
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue Sarcoma; Sarcoma,Soft Tissue; Sarcoma; Soft Tissue Sarcoma Adult
Keywords: soft tissue sarcoma; locally advanced soft tissue sarcoma; unresectable soft tissue sarcoma; metastasized soft tissue sarcoma; sarcoma; Retifanlimab; 20-316; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase I: Safety Run-In / Dose Level 0 (Experimental): A safety run-in (dose level 0 in Table 1, below) will be performed and enroll 6 patients with advanced high-grade sarcoma who are treatment naïve. Cycle one will consist of gemcitabine plus docetaxel at the institution's standard dose and schedule: 900 mg/m2 of gemcitabine on days 1 and 8, and 75 mg/m2 of docetaxel on day 8. Intravenous Retifanlimab at a flat dose of 210 mg will be administered every 3 weeks starting on C2D1 for a total of two cycles (cycles 2 and 3). All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Phase I: Dose De-escalation Level 1 (Experimental): If ≤ 1 patient out of 6 at dose level 0 has a dose-limiting toxicity during this safety run-in, then the dose de-escalation portion of the protocol will commence.
  Dose Level 1:
  Retifanlimab (Day 1) - 375 mg (flat dose) Gemcitabine (Days 1 and 8) - 900 mg/m2 Docetaxel (Day 8) - 75 mg/m2 All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Phase I: Dose De-escalation Level -1 (Experimental): Dose Level -1:
  Retifanlimab (Day 1) - 375 mg (flat dose) Gemcitabine (Days 1 and 8) - 750 mg/m2 Docetaxel (Day 8) - 60 mg/m2 All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Phase I: Dose De-escalation Level -2 (Experimental): Dose Level -2:
  Retifanlimab (Day 1) - 375 mg (flat dose) Gemcitabine (Days 1 and 8) - 675 mg/m2 Docetaxel (Day 8) - 50 mg/m2 All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Undifferentiated Pleomorphic Sarcoma/Myxofibrosarcoma (Experimental): (UPS/MFS)
  After the RP2D is determined, 5 histology-specific cohorts (10 patients each), including UPS/MFS, LPS, LMS, vascular sarcoma, and other STS, will open for enrollment. Patients will be treated with the RP2D of gemcitabine/docetaxel (when administered in combination with Retifanlimab) for cycle 1, with Retifanlimab added on cycle 2 day 1 at a flat dose of 375 mg. Gemcitabine/docetaxel will continue for 5 additional cycles (total of 6 cycles), after which treatment with Retifanlimab will continue until unacceptable toxicity, disease progression, or the completion of 35 cycles (105 weeks) of Retifanlimab treatment. All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Liposarcoma/LPS (Experimental): After the RP2D is determined, 5 histology-specific cohorts (10 patients each), including UPS/MFS, LPS, LMS, vascular sarcoma, and other STS, will open for enrollment. Patients will be treated with the RP2D of gemcitabine/docetaxel (when administered in combination with Retifanlimab) for cycle 1, with Retifanlimab added on cycle 2 day 1 at a flat dose of 375 mg. Gemcitabine/docetaxel will continue for 5 additional cycles (total of 6 cycles), after which treatment with Retifanlimab will continue until unacceptable toxicity, disease progression, or the completion of 35 cycles (105 weeks) of Retifanlimab treatment. All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Leiomyosarcoma/LMS (Experimental): After the RP2D is determined, 5 histology-specific cohorts (10 patients each), including UPS/MFS, LPS, LMS, vascular sarcoma, and other STS, will open for enrollment. Patients will be treated with the RP2D of gemcitabine/docetaxel (when administered in combination with Retifanlimab) for cycle 1, with Retifanlimab added on cycle 2 day 1 at a flat dose of 375 mg. Gemcitabine/docetaxel will continue for 5 additional cycles (total of 6 cycles), after which treatment with Retifanlimab will continue until unacceptable toxicity, disease progression, or the completion of 35 cycles (105 weeks) of Retifanlimab treatment. All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Vascular Sarcoma (Experimental): After the RP2D is determined, 5 histology-specific cohorts (10 patients each), including UPS/MFS, LPS, LMS, vascular sarcoma, and other STS, will open for enrollment. Patients will be treated with the RP2D of gemcitabine/docetaxel (when administered in combination with Retifanlimab) for cycle 1, with Retifanlimab added on cycle 2 day 1 at a flat dose of 375 mg. Gemcitabine/docetaxel will continue for 5 additional cycles (total of 6 cycles), after which treatment with Retifanlimab will continue until unacceptable toxicity, disease progression, or the completion of 35 cycles (105 weeks) of Retifanlimab treatment. All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Other Soft tissue sarcoma/STS (Experimental): After the RP2D is determined, 5 histology-specific cohorts (10 patients each), including UPS/MFS, LPS, LMS, vascular sarcoma, and other STS, will open for enrollment. Patients will be treated with the RP2D of gemcitabine/docetaxel (when administered in combination with Retifanlimab) for cycle 1, with Retifanlimab added on cycle 2 day 1 at a flat dose of 375 mg. Gemcitabine/docetaxel will continue for 5 additional cycles (total of 6 cycles), after which treatment with Retifanlimab will continue until unacceptable toxicity, disease progression, or the completion of 35 cycles (105 weeks) of Retifanlimab treatment. All visits are to be done +/-3 days of the scheduled timepoints.
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Docetaxel
- Advanced sarcoma who have progressed on prior treatment (Experimental): Participants will have advanced sarcoma who have progressed on prior treatment and have an immune-enriched/non-fibrotic TME
  Interventions: Drug: Retifanlimab

INTERVENTIONS:
Drug: Retifanlimab — Phase I:
  Dose Level 1 - 375 mg (flat dose) Dose Level 0 - 210 mg (flat dose) Dose Level -1 - 375 mg (flat dose) Dose Level -2 - 375 mg (flat dose)
  Phase II: 375 mg (flat dose)
  Other Names: INCMGA00012
Drug: Gemcitabine — Phase I:
  Dose Level 1 - 900 mg/m2 Dose Level 0 - 900 mg/m2 Dose Level -1 - 750 mg/m2 Dose Level -2 - 675 mg/m2
  The dose level with ≤ 1 DLT seen per patients will be declared the RP2D.
  Phase II: Participants will be treated with the RP2D of gemcitabine/docetaxel (when administered in combination with Retifanlimab ) for cycle 1, with Retifanlimab added on cycle 2 day 1 at a flat dose of 375mg. Gemcitabine/docetaxel will continue for 5 additional cycles (total of 6 cycles),
  Arms: Leiomyosarcoma/LMS; Liposarcoma/LPS; Other Soft tissue sarcoma/STS; Phase I: Dose De-escalation Level -1; Phase I: Dose De-escalation Level -2; Phase I: Dose De-escalation Level 1; Phase I: Safety Run-In / Dose Level 0; Undifferentiated Pleomorphic Sarcoma/Myxofibrosarcoma; Vascular Sarcoma
Drug: Docetaxel — Phase I:
  Dose Level 1 - 75 mg/m2 Dose Level 0 - 75 mg/m2 Dose Level -1 - 60 mg/m2 Dose Level -2 - 50 mg/m2
  The dose level with ≤ 1 DLT seen per patients will be declared the RP2D.
  Phase II: Participants will be treated with the RP2D of gemcitabine/docetaxel (when administered in combination with Retifanlimab) for cycle 1, with Retifanlimab added on cycle 2 day 1 at a flat dose of 375mg. Gemcitabine/docetaxel will continue for 5 additional cycles (total of 6 cycles),
  Arms: Leiomyosarcoma/LMS; Liposarcoma/LPS; Other Soft tissue sarcoma/STS; Phase I: Dose De-escalation Level -1; Phase I: Dose De-escalation Level -2; Phase I: Dose De-escalation Level 1; Phase I: Safety Run-In / Dose Level 0; Undifferentiated Pleomorphic Sarcoma/Myxofibrosarcoma; Vascular Sarcoma

SUMMARY:
This study is being done to find out whether the study drug Retifanlimab, a monoclonal antibody against the PD-1 protein, combined with gemcitabine and docetaxel, is a safe and effective treatment for your disease. Gemcitabine and docetaxel are chemotherapy drugs that are commonly used to treat soft tissue sarcoma. Retifanlimab is an experimental drug that boosts the immune system's ability to fight cancer cells. The study researchers think that Retifanlimab may help gemcitabine and docetaxel work better against soft tissue sarcoma that is either locally advanced or has spread beyond its original location (metastasized), and it cannot be removed with surgery (unresectable).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic or locally advanced and unresectable high-grade soft tissue sarcoma. Unresectable is defined as:

  1. primary tumor cannot be safely removed surgically, or
  2. primary tumor would benefit from systemic therapy prior to a surgical approach
* Be willing and able to provide written informed consent
* Must consent to mandatory tumor biopsy (if deemed safe and feasible) for research studies at screening, if archival tissue is not available, and at C1D15, C3D15.
* Age ≥ 18 years
* ECOG performance status ≤ 1
* Presence of measurable disease per RECIST v1.1

  * Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment.
* No prior systemic therapy (see exclusion criteria, below)
* Negative serum pregnancy test in women of childbearing potential
* Patients with chronic HBV (HBsAg-positive with undetectable or low HBV DNA and normal ALT, or HBsAg-negative with anti-HBc-positive serology) and HCV (completed curative antiviral treatment with HCV viral load below the limit of quantification) may be eligible

  * Patients with HBV should be treated with suppressive antiviral therapy prior to enrollment
  * Patients with HCV must have completed curative therapy and have negative HCV viral load
* Adequate organ function, as defined in Table 2:

Table 2: Laboratory Parameters Required for Study Inclusion

Hematological Absolute neutrophil count (ANC): ≥ 1,500 /mcL Platelets: ≥ 75,000 / mcL Hemoglobin: ≥ 9g/dL or ≥ 5.6 mmol/L

Renal Serum creatinine: ≤ 1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance: ≥ 60 mL/min for patient with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine orCrCl)

Hepatic Serum total bilirubin: ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN except patients with Gilbert's disease (≤ 3x ULN) AST (SGOT) and ALT (SGPT): ≤ 2.5 X ULN OR ≤ 5 X ULN for patients with liver metastases

Exclusion Criteria:

* Received any systemic therapy in the advanced or metastatic setting

  * Adjuvant or neoadjuvant therapies received ≥ 1 year prior to enrollment are permitted
* Unstable or deteriorating cardiovascular disease within the previous 6 months, including:

  * Unstable angina or myocardial infarction
  * CVA/stroke
  * New York Heart Association [NYHA] Class III or IV congestive heart failure
  * Uncontrolled clinically significant arrhythmias
* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment
* History or evidence of symptomatic autoimmune disease in past 2 years prior to enrollment.

  * Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease
* Uncontrolled HIV infection, as defined by one or more of the following:

  * Patients with CD4+ T-cell (CD4+) counts < 350 cells/uL
  * Patients with a history of an opportunistic infection secondary to AIDS
  * Patients on anti-microbials with drug-drug interactions with the study drugs on this protocol, who cannot be switched to alternative anti-microbials
  * Patients on antiretroviral therapy < 4 weeks
  * Patients with HIV viral load > 400 copies/mL
* Active Hepatitis B or Hepatitis C
* Patients who have received a live vaccine within 30 days of the start date of the planned study therapy (with the exception of COVID-19 vaccines)
* History of active TB (Bacillus Tuberculosis)
* Radiation therapy within 2 weeks prior to study day 1
* If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Women who are pregnant or breast feeding
* Patients expecting to conceive or father children within the projected duration of the trial, starting with the visit through 180 days after the last dose of study treatment(s)
* Prior organ transplantation including allogenic stem-cell transplantation
* Active infection requiring systemic therapy
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3)
* Patients with prior history of interstitial lung disease and clinically significant pulmonary compromise, including those who have a requirement for supplemental oxygen use to maintain adequate oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Phase II: proportion of patients that are progression-free at 24 weeks by RECIST v1.1 | 24 weeks
  The primary objective of the phase II portion of this study is to determine the proportion of patients that are progression-free at 24 weeks by RECIST v1.1. Progressive disease is declared when there is an increase in sum of target disease ≥ 20%, stable disease when the change is > -30% and ≤ 20%, partial response when there is a decrease in sum of target disease ≥ 30%, and complete response when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org